CLINICAL TRIAL: NCT03216681
Title: An Observational, Open Label, Post Marketing Study to Evaluate the Safety and Effectiveness of Hoat Huyet Nhat Nhat Compared With Gingko Biloba EGb761 (Tanakan 40mg) in Patients With Symptoms Related to the Insufficient Blood Supply to the Brain
Brief Title: Hoat Huyet Nhat Nhat Versus Tanakan for Treatment of Symptoms Related to the Insufficient Blood Supply to the Brain
Status: Completed | Type: Observational
Sponsor: Nhat Nhat Pharmaceutical Company (Industry)
Responsible Party: Sponsor
Other Study IDs: HHNN-01
Record Dates: First submitted 2017-07-09; First posted 2017-07-13 (Actual); Last update posted 2018-10-23 (Actual); Status verified 2017-07

CONDITIONS: Insufficient Blood Supply to the Brain
MeSH Terms: interventions — Ginkgo biloba extract

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hoat Huyet Nhat Nhat: Administered orally twice a day, 2 tablets each time, for 45 days.
  Interventions: Drug: Hoat Huyet Nhat Nhat
- Tanakan 40mg: Administered orally three times a day, one tablet each time, for 45 days.
  Interventions: Drug: Tanakan 40mg

INTERVENTIONS:
Drug: Hoat Huyet Nhat Nhat — Administered orally twice a day, 2 tablets each time, for 45 days.
  Groups: Hoat Huyet Nhat Nhat
Drug: Tanakan 40mg — Administered orally three times a day, 1 tablet each time, for 45 days.
  Groups: Tanakan 40mg

SUMMARY:
The purpose of this study is to evaluate the effectiveness of Hoat Huyet Nhat Nhat on the reduction of common symptoms related to the insufficient blood supply to the brain such as headache, vertigo, dizziness, sleep disorders and forgetfulness; compared with Gingko Biloba Egb761 (Tanakan) after 45 days of treatment

ELIGIBILITY:
Inclusion Criteria:

* Male and Female more than 18 year old.
* With at least one of the symptoms related to the insufficient blood supply to the brain scored more than 5 out 10, on the Visual Analog Scale.
* Patients who will be using either Hoat Huyet Nhat Nhat or Tanakan following doctor's prescription or by patients own decision.
* Sign the informed consent form

Exclusion Criteria:

* Use of any medications for treatment of the insufficient blood supply to the brain in the last 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female patients with symptoms related to the insufficient blood supply to the brain.
Sampling Method: Non-Probability Sample
Enrollment: 750 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-04-01 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
The percentage of patients with symptoms related to the insufficient blood supply to the brain recovered after 45 days of treatment as assessed by Symptom Improvement Likert Scale in Hoat Huyet Nhat Nhat and Tanakan 40mg group | 45 days

SECONDARY OUTCOMES:
Change From Baseline to 45 days of the severity of headache symptom in patients with symptoms related to the insufficient blood supply to the brain as assessed by Visual Analog Scale (VAS) | 45 days
Change From Baseline to 45 days of the severity of vertigo symptom in patients with symptoms related to the insufficient blood supply to the brain as assessed by Visual Analog Scale (VAS) | 45 days
Change From Baseline to 45 days of the severity of dizziness symptom in patients with symptoms related to the insufficient blood supply to the brain as assessed by Visual Analog Scale (VAS) | 45 days
Change From Baseline to 45 days of the severity of sleep disorders symptom in patients with symptoms related to the insufficient blood supply to the brain as assessed by Visual Analog Scale (VAS) | 45 days
Change From Baseline to 45 days of the severity of forgetfulness symptom in patients with symptoms related to the insufficient blood supply to the brain as assessed by Visual Analog Scale (VAS) | 45 days
Change From Baseline to 45 days of the severity of all symptoms related to the insufficient blood supply to the brain as assessed by Khadjev Score | 45 days
The number of participants with clinically significant vital sign parameters at Day 45. | 45 days
The number of participants with clinically significant laboratory parameters at Day 45. | 45 days

CONTACTS AND LOCATIONS:
Locations (1):
- Vietnam Military Medical University, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: Undecided